CLINICAL TRIAL: NCT04873583
Title: High Dose Steroids in Children With Stroke and Unilateral Focal Arteriopathy: A Multicentre Randomized Controlled Trial PASTA (Paediatric Arteriopathy Steroid Aspirin) Trial
Brief Title: High Dose Steroids in Children With Stroke
Acronym: PASTA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); LUMIS International GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1473_PASTA; 2022-500631-36-00 (EU CTIS Number); 2021-005571-39 (EudraCT Number); 2021-00453 (Other: Swissethics (BASEC Number)); 305395 (Other: HRA UK (IRAS Number)); HREC/78937/RCHM-2022 (Other: HREC Australia)
Record Dates: First submitted 2021-04-15; First posted 2021-05-05 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Paediatric Stroke
Keywords: Ischemic; Stroke; Pediatric; Steroids; Unilateral; Focal; Arteriopathy; Neurology; Cerebral
MeSH Terms: conditions — Ischemia; Stroke | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Prednisolone

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized, controlled, non-blinded trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Steroids + Standard of care (Experimental): Standard of care (including aspirin) and intravenous steroids, followed by oral tapering.
  Interventions: Drug: Methylprednisolone; Drug: Prednisolone
- Standard of care (No Intervention): Standard of care (including aspirin)

INTERVENTIONS:
Drug: Methylprednisolone — At the time of inclusion, intravenous Methylprednisolone for 3 days. Dose: 30 mg/kg/day (max. 1000 mg/dose)
  Other Names: Solu-Medrol
  Arms: Steroids + Standard of care
Drug: Prednisolone — Intravenous treatment will be immediately followed by oral tapering with Prednisolone.
  Oral Prednisolone, 2 weeks (week 1 and 2) Dose: 1 mg/kg/day (max 40 mg/day) Oral Prednisolone, 2 weeks (week 3 and 4) Dose: 0.5 mg/kg/day (max 20 mg/day)
  Other Names: Spiricort
  Arms: Steroids + Standard of care

SUMMARY:
This clinical trial deals with focal cerebral arteriopathy and childhood stroke, a rare but devastating condition.

Focal cerebral arteriopathy (FCA) is an inflammatory vessel wall disease provoked by infection and there is increasing evidence that inflammatory processes play a crucial role in childhood stroke, influencing the outcome of the disease.

Analysis of existing data suggests that outcomes are improved and that there is less stroke recurrence in children treated with steroids to reduce the acute inflammatory processes. This clinical trial will be conducted in over 20 hospitals in several countries in order to investigate this.

Participants will be randomly separated into two groups. The first group will be treated with standard of care (including aspirin) combined with high dose steroids. The second group will be treated with standard of care (including aspirin) but without steroid treatment.

The objective is to investigate if children treated with a combination of high dose steroid and aspirin will have a better and quicker recovery of FCA, better clinical functional outcome, and less recurrence compared to children treated with aspirin alone.

This project has been identified by international pediatric stroke experts as the most important topic for a clinical trial in the field and is as well one of the most important research priorities identified by parents. The study results will also provide insight into the evolution of inflammatory vessel disease.

DETAILED DESCRIPTION:
Background: Arterial ischemic stroke (AIS) is a rare but devastating condition affecting 2-5/100,000 children/year. Children do not recover better than adults with 2/3 suffering long term neurological, cognitive and behavioural problems. The economic cost of stroke is substantial. Arteriopathy is identified as AIS aetiology in 60-80% of previously healthy children and is the strongest predictor of recurrent events. 30-40% of these children will have a focal cerebral arteriopathy (FCA). FCA in childhood is shown to be an inflammatory vessel wall pathology provoked by infections. This encourages treatment with steroids, despite lack of evidence.

Rationale: There is increasing evidence that etiologically inflammatory processes play a crucial role in childhood stroke, and influence outcome. Retrospective analyses suggest improved outcome and less recurrence with steroid treatment. With the exception of sickle cell disease, this study will be the first randomized clinical trial in children with arterial ischemic stroke. It will provide high-level evidence for the most appropriate treatment for children with AIS due to FCA. Alignment of interventions and outcome as well as pooled analysis with the planned Focal Cerebral Arteriopathy Steroid (FOCAS) study in North America will allow pooled analysis results.This is very important in view of the marked neurological, social and economic burden of childhood AIS for patients and families. This project has been identified as the most important AIS treatment trial by a Delphi survey of international paediatric stroke experts and is one of the most important research priorities identified by parents. In addition, the study will provide insights into the pathogenesis of inflammatory vasculopathies.The objective of this trial is to show that children with first stroke event due to unilateral FCA treated with a combination of high dose steroid and aspirin will have better and quicker recovery of arteriopathy, better clinical functional outcome, and less recurrence compared to children treated with aspirin alone.

The proposed study is a prospective multicentre, parallel group, two-arm, randomized controlled, open-label clinical trial with blinded outcome assessment, comparing a high dose course of methylprednisolone / prednisolone plus standard of care with standard of care alone in children with unilateral arteriopathy and acute ischemic stroke.

Measurements and procedures: Participants will be randomized within 48 hours after diagnosis (maximum 96 hours after stroke onset) to standard of care (SC) alone (control group) or SC plus steroids (experimental group). SC will be harmonized among the study centres to include aspirin treatment. Patients will be assessed at 1, 3, 6 and 12 months. Magnetic imaging and angiography (MRI/MRA) will be done at 1, (3) and 6 months.

Number of Participants: 70 participants in total, 35 per treatment arm

Study duration: 48 months

Study Centre(s): International multi-centre study with approximately 20 to 30 centres

Participating countries:Switzerland, Germany, France, Austria, Great Britain & Australia

Centres in additional countries might be considered.

Statistical Considerations: The sample size is based on the comparison of the primary outcome - the change in FCASS from baseline to 1 month - between the two treatment groups. The standard deviation from 13 patients of a retrospective study was calculated. The standard deviation of the baseline and follow-up FCASS was 3.0 and 3.3, respectively. The standard deviation of the change in FCASS from baseline was 2.8. Based on the standard deviation of 2.8 and a two-sample means test, 64 patients (32 in each group) are required to detect a difference of 2.0 with a power of 80% at a two-sided alpha-level of 0.05. To account for dropouts (8%), we enlarge the sample size to 70 patients (35 in each group). The primary analysis will follow the intention-to-treat (ITT) principle, i.e. all patients will be analysed in the allocated group regardless of any protocol violations such as cross-overs. The primary outcome (change in FCASS from baseline to 1 month) as well as other secondary continuous score outcomes that are measured multiple times during follow-up (RRQ, mRS, Pediatric Stroke Outcome Measure (PSOM), VABS, modAspect) will be assessed in a repeated-measure, mixed-effects linear model.

Good Clinical Practice (GCP) Statement: This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH-GCP) as well as all national legal and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent of the legal representative of the trial participant documented by signature
2. Age > 6 months & < 18 years at time of stroke
3. Randomisation possible within 48 hours of diagnosis and maximum 96 hours after stroke onset
4. Unilateral arteriopathy according to the following criteria:

   * Newly acquired neurologic deficits
   * Specific neuroimaging (MRA) features of either

     * unilateral stenosis, or
     * unilateral vessel irregularities within the Central Nervous System (CNS)
5. Unless otherwise defined in the national addendum: Female participants age ≥ 13: Negative pregnancy test (blood or urine)

Exclusion Criteria:

1. Previous stroke
2. Known syndromal disorders, as e.g. Trisomy 21, Neurofibromatosis type 1
3. Known genetic vasculopathies as e.g. posterior fossa anomalies, hemangioma, arterial anomalies, cardiac anomalies and eye anomalies syndrome (PHACES), actin alpha 2 (ACTA II)
4. Moyamoya or sickle cell disease
5. Small vessel cerebral vasculitis (primary CNS vasculitis)
6. Bilateral arteriopathy
7. Arterial dissection(s)
8. Evidence of underlying systemic disorders, as e.g. lupus, rheumatoid problems
9. Secondary CNS angiitis due to infections (meningitis, endocarditis, borreliosis), or generalised angiitis due to rheumatic or other autoimmune problems
10. Progressive large to medium childhood primary angiitis of the CNS (cPACNS ) with 2 of the following 3 criteria:

    1. pre-existing progressive neurocognitive dysfunction
    2. bilateral MRI lesions/vessel involvement
    3. small vessel arterial stenosis
11. On steroid treatment at disease onset
12. Contraindication to steroid treatment as e.g. a congenital or acquired immunodeficiency
13. Inability to follow the procedures of the study, e.g. due to language problems
14. Participation in another interventional study within the 30 days preceding the indication stroke and during the present study

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Focal Cerebral Arteriopathy Severity Score (FCASS) from baseline | 1 month (30 days)
  The FCASS is a scaling system that has been developed to improve diagnostic criteria and to better document the typical course of initial worsening followed by improvement in FCA-i (focal cerebral arteriopathy of inflammatory type).
  FCASS Minimum score (best outcome): 0 FCASS Maximum baseline score (worst outcome): 20 FCASS Maximum follow up score (worst outcome): 21

SECONDARY OUTCOMES:
Functional impairment outcome measured by Pediatric Stroke Outcome Measure (PSOM) | 1, 3, 6 and 12 months
  The PSOM is a measure that has been specifically developed and validated for pediatric stroke patients and addresses pediatric specific domains such as development, behavior and cognition in addition to sensory-motor and language function.
  PSOM Minimum score (best outcome): 0 PSOM Maximum baseline score (worst outcome): 10
Recovery assessed by Recovery and Recurrence Questionnaire (RRQ) | 1, 3, 6, and 12 months
  The Pediatric Recovery and Recurrence Questionnaire was specifically developed and validated for pediatric stroke patients and addresses pediatric- specific problems of manifestation of stroke and difficulties in reliable clinical examination.
  Minimum score (best outcome): 0 Maximum baseline score (worst outcome): 10
Degree of disability or dependence by modified Rankin Scale (mRS) | 1, 3, 6, and 12 months
  Minimum score (best outcome): 0 Maximum baseline score (worst outcome): 6
Clinical outcome by Vineland adaptive behavior scale (VABS) | 6 and 12 months
  The vineland adaptive behavior scale is a validated instrument to monitor cognitive and behavior problems of children by interview.
  (range=40-160, the higher the score the better the performance)
Change in FCASS (Focal Cerebral Arteriopathy Severity Score) from baseline | 6 months
  The FCASS is a scaling system that has been developed to improve diagnostic criteria and to better document the typical course of initial worsening followed by improvement in FCA-i (focal cerebral arteriopathy of inflammatory type).
  FCASS Minimum score (best outcome): 0 FCASS Maximum baseline score (worst outcome): 20 FCASS Maximum follow up score (worst outcome): 21
Volume of stroke | baseline, 1, 3 (if imaging is available) and 6 months
  Volume of stroke will be measured by modASPECTS in diffusion-weighted MRI (DWI) and fluid-attenuated inversion recovery (FLAIR) images.
  Higher scores represent greater volumes, with a range of 0-30 (15 per hemisphere).
  modASPECTS: Modified pediatric ASPECTS
  ASPECTS: Alberta stroke program early CT score
Residual vasculopathy | 6 months
  Residual vasculopathy measured by FCASS (Focal Cerebral Arteriopathy Severity Score)
  The FCASS is a scaling system that has been developed to improve diagnostic criteria and to better document the typical course of initial worsening followed by improvement in FCA-i (focal cerebral arteriopathy of inflammatory type).
  FCASS Minimum score (best outcome): 0 FCASS Maximum baseline score (worst outcome): 20 FCASS Maximum follow up score (worst outcome): 21
Stroke recurrence after index stroke | 1, 6 and 12 months
  Stroke recurrence is defined as
  (i) new focal neurological deficit(s)
  (ii) worsening of the neurological deficits by > 4 pedNIHSS points lasting for more than 24 hours with new or increased diffusion restriction at the time of recurrence (with or without FLAIR/T2 lesions) in the corresponding vascular territory, or
  (iii) new areas of clinically silent infarction, remote from the initial infarct (at 1 and 6 months)
Stroke recurrence after index stroke in relation to the initial degree of vessel stenosis | 6 and 12 months
  Degree of vessel stenosis measured by change in FCASS from baseline to follow-up.
  Stroke recurrence will be measured as proportion in each category of vessel stenosis.
Stroke Quality of Life Measure (PSQLM) | 12 month
  For children between 2 -18 years quality of life will be assessed with the Pediatric Stroke Quality of Life Measure (PSQLM) (range=-10 to 10, the higher the score the better the performance)
Preschool Wechsler Intelligence Scale for Children (WISC V) / Wechsler Preschool and Primary Scale of Intelligence (WIPPSI IV) | 12 month
  For Children between 2 -18 years intelligence will be assessed by Preschool Wechsler Intelligence Scale for Children (WISC V) / Wechsler Preschool and Primary Scale of Intelligence (WIPPSI IV, as age appropriate) (range=40-160, the higher the score the better the performance)
Delis-Kaplan Executive Function System (D-KEFS) | 12 month
  Children > 8 years will undergo specific evaluation of executive function (EF). They will be assessed with the Delis-Kaplan Executive Function System (D-KEFS) Trail Making Test, Delis-Kaplan Executive Function System (D-KEFS) Color-Word-Interference Test (range=1-19, the higher the score the better the performance)
Continuous performance task (CPT-III) | 12 month
  Children > 8 years will undergo specific evaluation of attention. They will be assessed with the Continuous performance task (CPT-III). (range=20-80, the higher the score the better the performance)

CONTACTS AND LOCATIONS:
Overall Officials: Maja Steinlin, Prof. em. Dr. med., Study Director — Bern university hospital, Inselspital Bern, Kinderklinik
Locations (35):
- Australia (3):
  - Sydney Childrens Hospital Randwick, Randwick, New South Wales
  - Sydney Childrens Hospital Network, Westmead, New South Wales
  - Melbourne Childrens Hospital, Melbourne, Victoria
- Austria (3):
  - Universitätsklinik für Pädiatrie 1 A.ö. Landeskrankenhaus/ Universitätskliniken Innsbruck, Innsbruck, Tyrol
  - Johannes Kepler University Linz, Med Campus IV, Univ.-Klinik für Kinder- und Jugendheilkunde, Linz, Upper Austria
  - Universitätsklinik für Kinder und Jugendheilkunde Wien, Vienna
- Denmark (2):
  - Børn og Unge - Aarhus Universitetshospital, Aarhus
  - Department of Pediatric and Adolescence Medicine Copenhagen University Hospital, Copenhagen
- France (6):
  - L'ASSISTANCE PUBLIQUE-HOPITAUX DE MARSEILLE (AP-HM) - Hôpital de la Timone, Marseille, Aix-en-Provence
  - Pediatric Neurology Strasbourg - Hautepierre University Hospital, Strasbourg, Alsace
  - Hôpital Femme Mère Enfant Lyon, Bron, Auvergne-Rhône-Alpes
  - Hôpital Roger Salengro, CHRU de Lille, Lille
  - Hôpitaux Universitaires Paris Sud, Le Kremlin-Bicêtre, Île-de-France Region
  - Hôpital Necker-Enfants Malades, Paris, Île-de-France Region
- Germany (6):
  - Universitätsklinikum Freiburg Zentrum für Kinder- und Jugendmedizin Klinik für Neuropädiatrie und Muskelerkrankungen, Freiburg im Breisgau, Baden-Wurttemberg
  - LMU Klinikum, München, Bavaria
  - Universitätsklinikum Düsseldorf, Düsseldorf, Nordrhein-Westfahlen
  - Universitäts Kinderklinik Münster, Münster, Nordrhein-Westfahlen
  - Charité-Universitätsmedizin Berlin, Berlin
  - Medizinische Hochschule Hannover OE 6720, Hanover
- Centrum för Kliniska Barnstudier, Astrid Lindgrens Bansjukhus, Kaolinska Universitetssjukhuset, Stockholm, Sweden
- Switzerland (10):
  - Centre Hôpitalier Universitaire Vaud (CHUV), Unité de Neurologie, Lausanne, Canton of Vaud
  - Ospedale Regionale di Bellinzona e Valli, Bellinzona, Canton Ticino
  - Kantonsspital Graubünden, Departement Kinder- und Jugendmedizin, Chur, Kanton Graubünden
  - Hôpital du Valais, Sion, Valais
  - Universitätskinderklinik beider Basel, Basel
  - Inselspital Bern, Bern
  - Hôpitale Universitaire de Genève, Neuropediatrie, Hôpital des Enfants, Geneva
  - Luzerner Kantonsspital, Kinderspital, Neuropädiatrie, Lucerne
  - Stiftung ostschweizerisches Kinderspital, Sankt Gallen
  - Kidnerspital Zürich, Zurich
- United Kingdom (4):
  - Addenbrookes Hospital - Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire
  - University Hospital Southampton, Southampton, Hampshire
  - Royal Manchester Children's Hospital, Manchester, Lancashire
  - University Hospital Bristol, Bristol

IPD SHARING:
Plan to Share IPD: No
It is not planned to share individual participant data to other researchers.

REFERENCES:
- [Background] Steinlin M, O'callaghan F, Mackay MT. Planning interventional trials in childhood arterial ischaemic stroke using a Delphi consensus process. Dev Med Child Neurol. 2017 Jul;59(7):713-718. doi: 10.1111/dmcn.13393. Epub 2017 Jan 25. PMID 28121022
- [Derived] Fullerton HJ, Hills NK, Chen H, Dlamini N, Stence NV, Wintermark M; VIPS II Investigators. Changing Management of Focal Cerebral Arteriopathy of Childhood From 2010 to 2022. Stroke. 2025 Jun;56(6):1460-1468. doi: 10.1161/STROKEAHA.124.050550. Epub 2025 May 12. PMID 40351190
- See also: Protocol Publication — https://pediatricstrokejournal.com/high-dose-steroids-in-children-with-stroke-and-unilateral-focal-arteriopathy-a-multicenter-randomized-controlled-trial/